CLINICAL TRIAL: NCT03797274
Title: Quantitative Frontal Electroencephalography (EEG) and Postoperative Emergence Delirium Following General Anesthesia in Children: a Prospective Observational Study
Brief Title: Quantitative EEG During Anesthesia Emergence in Children
Acronym: qEEG
Status: Completed | Type: Observational
Sponsor: Daegu Catholic University Medical Center (Other)
Responsible Party: Principal Investigator, Eugene Kim, Assistant professor, Daegu Catholic University Medical Center
Other Study IDs: DCMC#7
Record Dates: First submitted 2019-01-05; First posted 2019-01-09 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Anesthesia, General; Electroencephalography; Brain Waves; Psychology, Children; Child Behavior
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Most drugs used in general anesthesia work on various receptors in the human brain, causing unconsciousness, loss of memory, and loss of reflection of the autonomic nervous system. After the anesthesia, baseline physiological function will be attained by administration of some reversal drugs or as the time goes by. In this process, various side effects may occur.

Emergence delirium (ED) is a representative behavioral disturbance after general anesthesia in children and that can cause several problems during the recovery period. Previous EEG studies reported that this phenomenon is related to hyperexcitation of the brain, and occurrence of epileptiform discharges during anesthesia induction may indicate an increased vulnerability for the development of a functional brain disorder in these children.

However, to the best of our knowledge, there is no studies concern evaluating quantitative EEG parameters for prediction of this postoperative negative behavior in children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 2 and 10 years of American Society of Anesthesiologists physical status (ASA PS) I or II who are planned to receive surgery under general anesthesia

Exclusion Criteria:

* If the guardian and the subject are difficult to evaluate normally due to language barriers/language disorders/delay or autistic disorder
* with developmental delay, neurological disorders or psychiatric diseases associated with symptoms of agitation, anxiety, attention deficit, sleep disturbances, etc
* refusal of consent
* Recent history (within a month) of received general anesthesia or surgery
* presence of congenital or other genetic conditions thought to influence brain development

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study collects subjects from a tertiary university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of Emergence delirium | During 60 minutes after PACU admission
  On arrival at post-anesthesia care unit (PACU), patients are checked post-anesthesia emergence delirium (PAED). The PAED scale is a validated observational measure of 5 aspects of child behavior (caregiver eye contact, purposeful movement, evidence of awareness of surroundings, restlessness, and inconsolability). Ratings are summed to produce a total score ranging from 0 to 20; greater scores indicate greater severity.
  If the PAED score is greater than 12, investigators define emergence delirium.
Relative power of each brain waves | From the cessation of sevoflurane inhalation to the extubation of airway devices such as tracheal tubes or laryngeal mask airway
  Original frontal EEG segments are attained via 2 channel bispectral index monitoring (BIS VISTA™, Aspect Medical Systems, Inc. MA, USA) during the anesthesia period. The EEG is then segmented into 4 s epochs and fast Fourier transform (FFT) analysis is performed for each of these segments. FFT of all these selected EEG segments are computed in the following frequency bands:
  Delta: 1-4 Hz Theta: 4-8 Hz Alpha: 8-13 Hz Beta: 13-30 Hz
  And then, the relative power of each frequency bands to the total power of the sum is calculated.

SECONDARY OUTCOMES:
modified Yale preoperative anxiety score (mYPAS) | before anesthesia induction (about 30 min before the surgery)
  mYPAS is the assessment tool for measure the anxiety before induction. Higher score indicates higher anxiety.
PAED score during PACU stay | During 60 min after PACU admission
  On arrival at post-anesthesia care unit (PACU) and every 10 min from then, patients were checked PAED. The PAED scale is a validated observational measure of 5 aspects of child behavior (caregiver eye contact, purposeful movement, evidence of awareness of surroundings, restlessness, and inconsolability). Ratings are summed to produce a total score ranging from 0 to 20; greater scores indicate greater severity.
FLACC score on initial, 10, 20, and 30 min | During 60 minutes after PACU admission]
  Face, legs, activity, cry, and consolability (FLACC) score is checked every 10min after PACU admission
Watcha scale on initial, 10, 20, and 30 min | During 60 minutes after PACU admission
  On arrival and 10, 20, and 30 min after PACU admission, patients were checked Watcha scale as following 4-point scale
  1. calm
  2. crying, but can be consoled
  3. Crying, cannot be consoled
  4. Agitated and thrashing around
  Higher score indicates higher agitation.
Delta-theta to alpha-beta ratio (DTABR) | From the cessation of sevoflurane inhalation to the extubation of airway devices such as tracheal tubes or laryngeal mask airway
  From the relative power of each brain waves, the investigators calculated the ratio as follows:
  DTABR = (Delta wave + Theta wave)/(alpha wave + beta wave)
Delta to alpha ratio | From the cessation of sevoflurane inhalation to the extubation of airway devices such as tracheal tubes or laryngeal mask airway
  From the relative power of each brain waves, the investigators calculated the ratio as follows:
  DAR = Delta wave / alpha wave
Theta to beta ratio (TBR) | From the cessation of sevoflurane inhalation to the extubation of airway devices such as tracheal tubes or laryngeal mask airway
  From the relative power of each brain waves, the investigators calculated the ratio as follows:
  TBR = Theta wave / beta wave

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Kim, MD, PhD, Study Chair — Assistant professor
Locations (1):
- Eugene Kim, Daegu, Nam-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim J, Lee HC, Byun SH, Lim H, Lee M, Choung Y, Kim E. Frontal electroencephalogram activity during emergence from general anaesthesia in children with and without emergence delirium. Br J Anaesth. 2021 Jan;126(1):293-303. doi: 10.1016/j.bja.2020.07.060. Epub 2020 Oct 1. PMID 33010926